CLINICAL TRIAL: NCT04960748
Title: Pilot of a Network-driven, Advocacy Intervention to Promote Cervical Cancer Screening in Uganda
Brief Title: Promoting Cervical Cancer Screening Through the Advocacy of Screened Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Makerere University (Other); Rays of Hope Hospice Jinja (Unknown); African Palliative Care Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21TW011728 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cervical Cancer Prevention
Keywords: cervical cancer screening; prevention advocacy; group intervention; Uganda; social networks

STUDY DESIGN:
Intervention Model Description: randomized controlled trial of parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): 7-sesson group intervention that uses dyadic instruction, role playing and group sharing and discussion to reduce internalized stigma, improve disclosure decision making and healthy living, and teach advocacy skills
  Interventions: Behavioral: WOMEN FIGHTING TO STOP CERVICAL CANCER
- wait-list control (No Intervention): Participants will not receive the intervention until all follow-up data has been collected.

INTERVENTIONS:
Behavioral: WOMEN FIGHTING TO STOP CERVICAL CANCER — The group intervention draws on theories of social diffusion, cognitive consistency, and social influence, and our own recently developed and tested group intervention that mobilized people living with HIV in Uganda to successfully act as change agents for HIV prevention within their social networks. The intervention actively targets internalized stigma, disclosure decision making, healthy living, and advocacy communication skills. The ultimate goal of the program is to encourage female social network members to get screened for cervical cancer.
  Arms: intervention

SUMMARY:
This study pilots a 7-session group intervention among 40 screened women, 20 of whom will be randomly assigned to take part in the intervention, and 20 to the wait-list control. Assessments will be administered at baseline and month 6 to index participants as well as up to three unscreened female social network members of each index participant (up to 120 total). The primary outcome is CC screening among participating social network members.

DETAILED DESCRIPTION:
Cervical cancer (CC) is the most common cancer and accounts for ~25% of all cancer related deaths among women in Uganda, which has one of the highest incidence rates in the world. Adding to the burden is the general lack of knowledge about, and social stigma towards CC and its screening in Uganda, where lifetime CC screening is estimated to be as low as 5%. There is a dire need to increase CC screening in Uganda to ensure timely and lifesaving treatment, as well as the need to enhance the capacity to conduct behavioral and health services research related to CC and other stigmatizing conditions among local researchers and service providers. Accordingly, the proposed intervention pilot study seeks to (1) empower women who have been screened for CC, to advocate for CC screening and early treatment among women in their social networks, and (2) engage and train local public health researchers and programmers. The proposed intervention draws on theories of social diffusion, cognitive consistency, and social influence, and the investigator's recently developed and tested group intervention that mobilized people living with HIV in Uganda to successfully act as change agents for HIV prevention within their social networks. The intervention actively targets internalized stigma, disclosure decision making, healthy living, and advocacy communication skills. This study will pilot the intervention among 40 screened women, 20 of whom will be randomly assigned to take part in the intervention, and 20 to the wait-list control. Assessments will be administered at baseline and month 6 to index participants as well as up to three unscreened female social network members of each index participant (up to 120 total). The primary outcome is CC screening among participating social network members. The primary aims of the study are to assess the feasibility, acceptability and preliminary efficacy of the group intervention to promote CC screening and treatment; identify characteristics associated with successful advocacy; and increase local capacity for conducting public health research on CC control and use of social network-based intervention and measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* has been previously screened for cervical cancer
* has told at least one woman in her social network about her cervical cancer screening experience

Exclusion Criteria:

* unstable medical status (e.g., advance disease stage that calls into question her ability to complete the 6-month study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — persons with female sex organs
Enrollment: 143 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Proportion of social network members who report cervical cancer screening | past 6 months
  cervical cancer screening among women in social network

SECONDARY OUTCOMES:
Proportion of index participants who self-report engagement in cervical cancer (CC) prevention advocacy | past 6 months
  discussing cervical cancer and encouraging CC screening with women in social network

CONTACTS AND LOCATIONS:
Overall Officials: Rhoda Wanyenze, MD, Principal Investigator — Makerere University
Locations (1):
- Buyinja HCIV, Namayingo, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wagner GJ, Matovu JKB, Juncker M, Namisango E, Bouskill K, Nakami S, Beyeza-Kashesya J, Luyirika E, Bogart LM, Green HD, Wanyenze RK. Effects of a peer advocacy intervention on cervical cancer screening among social network members: results of a randomized controlled trial in Uganda. J Behav Med. 2023 Dec;46(6):930-939. doi: 10.1007/s10865-023-00418-6. Epub 2023 Sep 13. PMID 37702912
- [Derived] Ghai I, Wagner GJ, Matovu JKB, Juncker M, Namisango E, Bouskill K, Nakami S, Beyeza-Kashesya J, Luyirika E, Wanyenze RK. Increased Knowledge Mediates the Effect of Game Changers for Cervical Cancer Prevention on Diffusion of Cervical Cancer Screening Advocacy Among Social Network Members in a Pilot Trial. Int J Behav Med. 2024 Oct;31(5):753-763. doi: 10.1007/s12529-023-10217-7. Epub 2023 Sep 1. PMID 37656308
- [Derived] Wanyenze RK, Matovu JKB, Bouskill K, Juncker M, Namisango E, Nakami S, Beyeza-Kashesya J, Luyirika E, Wagner GJ. Social network-based group intervention to promote uptake of cervical cancer screening in Uganda: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Dec 7;8(1):247. doi: 10.1186/s40814-022-01211-z. PMID 36476609